CLINICAL TRIAL: NCT01570309
Title: The Effects of Vitamin D Repletion on Endothelial Function and Inflammation in Patients With Coronary Artery Disease
Brief Title: Vitamin D Repletion in Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seth I. Sokol, M.D. (Other)
Collaborators: American Heart Association (Other); Jacobi Medical Center (Other); Albert Einstein College of Medicine (Other); Yale University (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor-Investigator, Seth I. Sokol, M.D., Principal Investigator, New York City Health and Hospitals Corporation
Organization: New York City Health and Hospitals Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHA Award #0885041N
Record Dates: First submitted 2012-03-26; First posted 2012-04-04 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-08

CONDITIONS: Vitamin D Deficiency; Coronary Artery Disease; Endothelial Dysfunction; Inflammation
Keywords: vitamin D,; vitamin D deficiency; coronary artery disease; ergocalciferol; endothelial function; adhesion molecules; inflammation; IL-12; interferon-gamma; CXCL-10; reactive hyperemia peripheral arterial tonometry; endothelial dysfunction; cytokines; chemokines
MeSH Terms: conditions — Vitamin D Deficiency; Coronary Artery Disease; Inflammation | interventions — Ergocalciferols; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ergocalciferol (Active Comparator): 50,000 units of ergocalciferol once a week for 12 weeks
  Interventions: Drug: Ergocalciferol
- Sugar pill (Placebo Comparator)
  Interventions: Other: Sugar pill

INTERVENTIONS:
Drug: Ergocalciferol — Oral capsule, 50,000 units, once a week, 12 weeks
  Arms: Ergocalciferol
Other: Sugar pill — Oral capsule, once a week, 12 weeks
  Arms: Sugar pill

SUMMARY:
Vitamin D (Vit D) status is an emerging risk marker of great interest in cardiovascular disease (CVD). Lower serum levels of Vit D are associated with both cardiac risk factors and prevalent cardiovascular disease. Vit D insufficiency remains very prevalent in free living populations in the United States especially in urban, and multi-ethnic low income Northern cities.To date, prospective randomized trials using Vit D supplementation to modify CVD risk and evaluate outcomes have not been performed.

The investigators propose a double-blind, randomized wait-list control trial in subjects with Coronary Artery Disease (CAD) and Vit D deficiency with two specific aims. Specific aim 1 is to measure endothelial function using reactive hyperemia peripheral arterial tonometry (RH-PAT) before and after treatment with Vit D replacement therapy. Specific Aim 2 is to measure levels of inflammation before and after treatment with Vit D replacement therapy. These aims will test the hypotheses that Vit D repletion will improve endothelial function and reduce the levels of detectable inflammation in the plasma of these subjects.

DETAILED DESCRIPTION:
100 subjects with angiographically documented CAD and Vit D deficiency will be randomized to 50,000 IU oral ergocalciferol (active treatment group) or placebo (delayed intervention group) once a week for 12 weeks. The investigators will measure endothelial function at randomization and week 12 using RH-PAT and serologically measured adhesion molecules (s-VCAM, s-ICAM, soluble e-selectin). Changes in levels of plasma cytokines and chemokines representing a T-cell activation pathway (IL-12, IFN-g and CXCL-10 - "IFN-g axis") the investigators have linked to coronary atherogenesis (independent of CRP) and poor CV outcomes, will be measured over the 12 week study period. Given published evidence showing that Vit D can influence this T- cell pathway, specific aim 2 will add mechanistic insights to this proposal. High sensitivity C-reactive protein (hs-CRP) will be measured as it is a well established traditional marker of inflammation in CAD and has also been linked to Vit D status.

ELIGIBILITY:
Inclusion Criteria:

* Male and nonpregnant females greater than 18 years of age
* ≥ 50% angiographic stenosis of at least 1 coronary artery or documented previous revascularization
* Serum 25-hydroxyvitamin D < 20 ng/ml

Exclusion Criteria:

* confinement to a nursing facility, institution or home
* GFR < 60 ml/min (by MDRD equation)
* presence of liver disease
* hypercalcemia
* NYHA class III or IV heart failure
* cardiogenic shock at time of presentation
* current planned or emergent CABG
* prior gastric or small bowel surgery
* pancreatitis
* malabsorption
* inflammatory bowel disease
* autoimmune disease
* active malignancy
* current use of > 800 IU/day of vitamin D
* Current use of dilantin, phenobarbitol, immunosuppressant, or immunostimulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth I Sokol, MD, Principal Investigator — Jacobi Medical Center
Locations (2):
- United States (2):
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center / Weiler division, The Bronx, New York

REFERENCES:
- [Result] Sokol SI, Srinivas V, Crandall JP, Kim M, Tellides G, Lebastchi AH, Yu Y, Gupta AK, Alderman MH. The effects of vitamin D repletion on endothelial function and inflammation in patients with coronary artery disease. Vasc Med. 2012 Dec;17(6):394-404. doi: 10.1177/1358863X12466709. PMID 23184900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from October 2008 through December 2010 from the cardiac catheterization laboratories and outpatient clinics of the Jacobi Medical Center and Montefiore Medical Center in the Northeastern section of the Bronx, NY. Additional recruitment occurred at Crystal Run Health in Orange County, NY.
Pre-assignment Details: Subjects with ≥ 50% angiographic stenosis of at least 1 coronary artery or documented previous revascularization, were screened for vitamin D deficiency by measurement of serum 25-hydroxyvitamin D (25-vitamin D).Eligible subjects with a 25-vitamin D level < 20 ng/ml were randomly assigned 1:1 to active or placebo treatment
Groups:
- Sugar Pill: Matching placebo
Period: Overall Study
Arm/Group | Ergocalciferol | Sugar Pill
Started | 48 | 48
Completed | 45 | 45
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ergocalciferol | Sugar Pill | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 35 | 78
  >=65 years | 5 | 13 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 54.6 (9.5) | 56.5 (11.7) | 55.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 39 | 33 | 72
Region of Enrollment [Number; unit: participants]
  United States | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Function
Description: Endothelial function was measured using peripheral arterial tonometry expressed as the reactive hyperemia index. The index is derived from the ratio of the post-to-pre occlusion peripheral arterial tonometry signal amplitude of the tested arm, divided by the post -to-pre occlusion ratio of the control arm. Median within subject change in endothelial function as measured by reactive hyperemia peripheral arterial tonometry index in each group is presented.
Time Frame: Baseline and 12 weeks
Population: Assuming a standard deviation of 0.6 in the change in RH-PAT score from baseline to 12 weeks, we estimated that the study would need a sample size of 45 patients per treatment group to have 80% power at a two tailed alpha=0.05 level to detect a minimum difference in change in RH-PAT score of 0.36 between treatment groups.
Measure: Median (Inter-Quartile Range); unit: reactive hypermia index
Arm/Group | Ergocalciferol | Sugar Pill
Number analyzed (Participants) | 45 | 45
reactive hypermia index | 0.13 [-0.235 to 0.495] | -0.04 [-0.355 to 0.275]

2. Primary Outcome: Inflammation -
Description: Median within subject change in hs-CRP levels between baseline and week 12 in active and placebo groups
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dl
Groups:
- Active: Ergocalciferal 50,000 U qweekly x 12 weeks
Arm/Group | Active | Sugar Pill
Number analyzed (Participants) | 45 | 45
mg/dl | -0.17 [-1.82 to 1.48] | -0.05 [-0.96 to 0.86]

3. Primary Outcome: Inflammation
Description: Median within subject change in interferon-gamma levels between baseline and week 12 in active and placebo groups
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Ergocalciferol | Sugar Pill
Number analyzed (Participants) | 45 | 45
pg/ml | -2.29 [-13.34 to 8.76] | -2.8 [-8.78 to 3.18]

4. Primary Outcome: Inflammation
Description: Median within subject change in cxcl-10 .levels between baseline and week 12 in active and placebo groups
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- Active Therapy: Ergocalciferol 50,000 U q weekly x 12 weeks
- Placebo: Sugar Pill
Arm/Group | Active Therapy | Placebo
Number analyzed (Participants) | 45 | 45
pg/ml | -7.45 [-27.35 to 12.45] | -2.72 [-15.12 to 9.68]

5. Primary Outcome: Inflammation
Description: Median within subject change in IL-12 levels between baseline and week 12 in active and placebo groups
Time Frame: Baseline to week 12
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Ergocalciferol | Sugar Pill
Number analyzed (Participants) | 45 | 45
pg/ml | -10.96 [-43.46 to 21.54] | -2.33 [-27.18 to 22.52]

ADVERSE EVENTS:
Arm/Group | Ergocalciferol | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 10/45 | 9/45
Other Adverse Events (participants affected / at risk) | 4/45 | 4/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ergocalciferol (N=45) | Sugar Pill (N=45)
Death (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure exacerbation (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ICD shock inappropriate (Cardiac disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Angina (Cardiac disorders) | 0 (0) | 3 (3)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Atypical chest pain (Cardiac disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ergocalciferol (N=45) | Sugar Pill (N=45)
Headache (General disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No